CLINICAL TRIAL: NCT01338766
Title: Spondylolisthesis Treated With an iO-Flex® System Enabled Decompression (STRiDE)
Brief Title: Spondylolisthesis Treated With an iO-Flex® System Enabled Decompression
Acronym: STRiDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baxano Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-1967
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Radiculopathy; Spondylolisthesis; Lumbar Spinal Stenosis
Keywords: spondylolisthesis; lumbar spinal stenosis
MeSH Terms: conditions — Radiculopathy; Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): Decompression using the iO-Flex® system
  Interventions: Procedure: Decompression using the iO-Flex® system

INTERVENTIONS:
Procedure: Decompression using the iO-Flex® system — Decompression using the iO-Flex® system

SUMMARY:
The purpose of this study is to evaluate the clinical performance of a decompression using the FDA cleared iO-Flex® System on-label in treating patients with spinal stenosis and stable grade I degenerative lumbar spondylolisthesis using a precision estimate assuming a 55% positive response rate.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center (up to 30 sites) controlled clinical study enrolling 100 subjects following a pre-specified protocol with no site enrolling more than 30 subjects. All eligible subjects providing written informed consent and meeting study eligibility criteria will receive a facet preserving decompression using the FDA cleared iO-Flex® system on label. Treatment success using the iO-Flex® System will be analyzed using a precision estimate assuming a 55% positive response rate.

In addition to baseline characteristics and procedural parameters, subject outcomes will be assessed at 6 weeks, 6-, 12-, and 24 months. The study will have an extended follow-up phase with annual follow-up contact through 5 years to evaluate retreatment for the original indication at these late time points.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (> 18 years of age)
2. Leg/buttock pain, with or without back pain
3. Grade 1 degenerative spondylolisthesis (≤25% slippage)
4. NRS pain score for leg pain of 4/10 or greater
5. ODI score of 30/100 or greater
6. Failed non-operative medical management for a period of at least 6 months
7. Confirmed clinical diagnosis of lumbar spinal stenosis
8. Confirmation of central and/or lateral recess stenosis with or without foraminal stenosis, at one level or at two adjacent levels from L2-S1, with concordant symptoms. Subjects with central and/or lateral recess stenosis and spondylolisthesis at one level, may have symptomatic central, lateral recess or foraminal stenosis treated at one adjacent level. A "below-the pedicle" pass to decompress a third segment can be completed provided laminotomies are performed at no more than 2 levels. Subjects that, following an intraoperative decision, have a 3-level laminotomy and decompression will not be considered enrolled. Confirmation of spinal stenosis is shown on MRI or CT scan with evidence of nerve root impingement (displacement or compression) by either osseous or non-osseous elements.
9. Ability to give voluntary, written informed consent to participate in this clinical investigation and ability to participate in follow up examinations and complete patient questionnaires

Exclusion Criteria:

1. Back pain only
2. Diagnosis of moderate to severe peripheral neuropathy such as diabetic or idiopathic peripheral neuropathy, by EMG/NCS or a Neurologist.
3. History of pathologic fractures of the vertebrae
4. Primary disc pathology; planned or incidental discectomies will NOT be excluded as long as surgeon believes the disc pathology is not the primary reason for the surgical intervention.
5. Subjects for whom removal of the midline structures is planned, likely or is the result of an intraoperative decision; every attempt should be made to spare the supraspinous, interspinous and facet capsular ligaments.
6. Significant instability of the lumbar spine as defined by ≥ 4mm translational motion between standing lateral view flexion and extension radiographs
7. Prior surgery of the lumbar spine
8. Spondylolisthesis greater than grade 1 (on a scale of 1 to 4)
9. Spondylolysis (pars fracture) at any level in the lumbar spine
10. Degenerative lumbar scoliosis with a Cobb angle of ≥ 25°
11. Vascular claudication in the lower extremities
12. Cauda equina syndrome
13. Evidence of active (systemic or local) infection at time of surgery
14. Paget's disease at involved segment or metastasis to the vertebra, osteomalacia, or other metabolic bone disease
15. Tumor in the spine or a malignant tumor except for basal cell carcinoma.
16. Prisoner or transient
17. Any significant psychological disturbance past or present, psychotic or neurotic that could impair the consent process or ability to complete subject self-report questionnaires
18. Involved in pending litigation of the spine or worker's compensation related to the back
19. Inability to communicate clearly in the English language
20. Morbid obesity (BMI > 40)
21. Pregnant, nursing, or planning on becoming pregnant.
22. History of narcotic abuse
23. Current involvement in another drug or device clinical trial
24. Uncontrolled diabetes
25. Irreversible coagulopathy or bleeding disorder (patients on anticoagulant therapy may participate. Investigators should follow routine practices for perioperative discontinuation and reinitiation of anticoagulants.)
26. Plans to relocate in the next 2 years
27. Subject unwilling to undergo a blood transfusion, if necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 24 Months
  Responder analysis

SECONDARY OUTCOMES:
Operative success | Operative (day 1)
  Achieving intended decompression using the iO-Flex® System. The number of neural foramen in which the iO-Flex® System was used for decompression compared to the number in which an attempt was made but not completed.
Oswestry Disability Index (ODI) | 6, 12, 36, 48 and 60 months
  Responder analysis
Oswestry Disability Index (ODI) | 6, 12, 24, 36, 48 and 60 months
  Comparison of ODI scores between baseline and each of the following follow-up visits: 6, 12, 24, 36, 48, and 60 month visits
Numerical Rating Scale (NRS) | 6, 12, 24, 36, 48 and 60 months
  Comparison of NRS scores for back and leg pain between baseline and each of the following follow-up visits: 6, 12, 24, 36, 48, and 60 month visits
Zurich Claudication Questionnaire (ZCQ) | 6, 12, 24, 36, 48 and 60 months
  Comparison of ZCQ scores between baseline and each of the following follow-up visits: 6, 12, 24, 36, 48, and 60 month visits
SF-36 Health Survey | 6, 12, 24, 36, 48 and 60 months
  Comparison of SF-36 scores between baseline and each of the following follow-up visits: 6, 12, 24, 36, 48, and 60 month visits
Treatment survival rate | Ongoing out to 60 months
  To characterize longevity of the treatment effect of a decompression using the iO-Flex® System.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Palmer, M.D., Principal Investigator — Neurological Surgery Medical Associates
Locations (14):
- United States (14):
  - Eden Medical Center, Castro Valley, California
  - Olympia Medical Center, Los Angeles, California
  - Orange County Neurological Associates, Mission Viejo, California
  - University California Irvine, Orange, California
  - Southern California Orthopedic Institute, Van Nuys, California
  - Georgetown University, Washington D.C., District of Columbia
  - Medical Center of Trinity, Odessa, Florida
  - Florida Orthopaedic Institute, Temple Terrace, Florida
  - Resurgens Orthopaedics, Cumming, Georgia
  - Suburban Orthopedics, Bartlett, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Scott and White Memorial Hospital, Temple, Texas
  - VCU Medical Center, Richmond, Virginia
  - Tuckahoe Orthopedics, Richmond, Virginia